CLINICAL TRIAL: NCT04100473
Title: A Randomized, Open-Label, 6-Period Cross-Over Study to Investigate the Dose Response of Dance 501 (Human Insulin Inhalation Solution and Inhaler) in Subjects With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Dose Response of Dance 501 in Subjects With Type 2 Diabetes Mellitus
Acronym: T2DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dance Biopharm Inc. (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Samba-04
Record Dates: First submitted 2019-02-25; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Inhaled Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, Cross-Over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dance 501 (Experimental): Dance 501(Human Insulin Inhalation Solution and Inhaler) will be administered using the Dance 501 Inhaler.
  Interventions: Drug: Inhaled Human Insulin
- Insulin Lispro (Active Comparator): Insulin Lispro (Humalog®) will be administered by subcutaneous injection.
  Interventions: Drug: Insulin Lispro (Humalog U-100)

INTERVENTIONS:
Drug: Inhaled Human Insulin — Dance 501 administered using the Dance 501 Inhaler
  Other Names: Dance 501
  Arms: Dance 501
Drug: Insulin Lispro (Humalog U-100) — Lispro
  Other Names: Insulin Lispro (Humalog U-100) will be administered by subcutaneous injection
  Arms: Insulin Lispro

SUMMARY:
This will be a randomized, open-label, active-controlled, 6-period crossover study. Target population will be subjects with Type 2 Diabetes Mellitus (T2DM)

DETAILED DESCRIPTION:
To assess the dose-response and dose-exposure of Dance 501 (Human Insulin Inhalation Solution) administered with the Dance 501 Inhaler.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with T2DM.
* BMI between 25.0 and 40.0 kg/m2.
* Treated with metformin and/or at least 1 daily injection of insulin for at least 6 months.
* Non-smoker for at least 5 years.
* Forced vital capacity and forced expiratory volume in one second is at least 75% normal.

Exclusion Criteria:

* Any condition affecting pulmonary drug absorption.
* History or presence of cancer except basal cell skin cancer or squamous cell skin cancer.
* Serious systemic infectious disease during four weeks prior to dosing.
* Clinically significant abnormal lab values.
* Proliferative retinopathy and/or severe neuropathy.
* Recurrent severe hypoglycemia.
* Current treatment with oral anti-diabetic drugs except metformin, glucagon-like peptide receptor agonists.
* Current treatment with MAO inhibitors.
* Unstable Thyroid hormones for at least 3 months.
* Insufficient glycemic control with significant fluctuations of blood glucose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Primary Pharmacokinetic Endpoint - PK 1 | 0 - 10 hours
  Area under the human insulin and insulin lispro concentrations time curves
Primary Pharmacokinetic Endpoint - PK 2 | 0 - 10 hours
  Maximum observed concentration of human insulin and insulin lispro
Primary Pharmacodynamic Endpoint - PD 1 | 0 - 10 hours
  Area under the glucose infusion rate time curve
Primary Pharmacodynamic Endpoint - PD 2 | 0 - 10 hours
  Maximum observed glucose infusion rate

SECONDARY OUTCOMES:
Secondary Pharmacokinetic Endpoint - PK 1 | 0 - 1 hour, 0 - 2 hours, 0 - 8 hours
  Area under the insulin time curves at different intervals
Secondary Pharmacokinetic Endpoint - PK 2 | 0 - 10 hours
  Time to maximum insulin concentrations
Secondary Pharmacokinetic Endpoint - PK 3 | 0 - 10 hours
  Relative Efficiency of dose corrected ratio of AUC ins for INH and s.c. lispro
Secondary Pharmacokinetic Endpoint - PK 4 | 0 - 10 hours
  Onset of appearance (time from trial product administration until the serum insulin concentrations are > LLOQ.
Secondary Pharmacokinetic Endpoint - PK 5 | 0 - 10 hours
  Mean residence time of insulin
Secondary Pharmacodynamic Endpoint - PD 1 | 0 - 1 hour, 0 - 2 hours, 0 - 8 hours
  AUC for GIR at different time intervals
Secondary Pharmacodynamic Endpoint - PD2 | 0 - 10 hours
  Time to maximum glucose infusion rate
Secondary Pharmacodynamic Endpoint - PD3 | 0 - 10 hours
  Relative biopotency of dose corrected ratio of AUC GIR for INH and s.c. lispro

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Klein, Principal Investigator — Profil Institut fur Stoffwechselforschung GmbH
Locations (1):
- Profil Mainz, Mainz, Malakoff-Passage, Germany

IPD SHARING:
Plan to Share IPD: No